CLINICAL TRIAL: NCT00788996
Title: Effectiveness of a Brief Intervention Opportunistic Targeting Parents Who Smoke to Reduce Exposure to Secondhand Smoke in Babies: STUDY BIBE
Brief Title: Reduction of Environmental Tobacco Smoke (ETS) Exposure at Home: the BIBE Study
Acronym: BIBE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Comité Nacional Prevención Tabaquismo (Unknown); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other); Unitat Suport Recerca Àmbit Atenció Primària Barcelona. Institut Català Salut (Unknown)
Responsible Party: Guadalupe Ortega, Catalan Society of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNPT0701
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Tobacco Smoke Pollution
Keywords: Tobacco Smoke Pollution/prevention and control; Parent-Child Relations; Environmental Tobacco Smoke (ETS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Usual care
  Interventions: Behavioral: Brief intervention based in clinical practice guide

INTERVENTIONS:
Behavioral: Brief intervention based in clinical practice guide — Minimal counseling at smoking parents with babies minor 1 year-old
  Other Names: Usual care

SUMMARY:
Main objective: to determine the effectiveness of a brief opportunist educational performance directed to the parents who smoke -- inside the context of programmed visits of paediatrics in primary care -- to reduce the exposure of the babies to secondhand smoke (SHS)

Secondary objectives:

1. Smoking reduction / quitting of the mother and/or the father
2. To determine the relationship between the level exposure to SHS and main related variables

ELIGIBILITY:
Inclusion Criteria:

* Smoking parents with babies minor 1 year-old

Exclusion Criteria:

* Parents reporting diagnosis of major psychiatric illnesses
* Parents reporting active addictive substances consumption
* Parents in active smoking cessation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
The level of exposure to SHS in the babies by means of questionnaire and nicotine hair analysis. | 6 months at the beginning of intervention

SECONDARY OUTCOMES:
Parental smoking quitting or reduction by questionnaire and CO monitoring to whom self declared abstinent. Health related variables of babies and parents by follow-up questionnaire | 6 months at the beginning of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ortega Guadalupe, Nurse, Principal Investigator — Direcció General de Salut Pública. Departament de Salut. Catalunya
Locations (1):
- Direcció General de Salut Pública, Departament de Salut, Catalunya, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Ortega Cuelva G, Cabezas Pena C, Almeda Ortega J, Saez Zafra M, Ballve Moreno JL, Pascual Esteban JA, Castella Cuesta C, Martin-Cantera C, Salto Cerezuela E, Casademont Pou RM, Diaz Alvarez E, Lozano Fernandez J, Morera Jordan C, Valverde Trillo A, Perez-Ortuno R, Rofes Ponce L, Jane Checa M; BIBE study group. Effectiveness of a brief primary care intervention to reduce passive smoking in babies: a cluster randomised clinical trial. J Epidemiol Community Health. 2015 Mar;69(3):249-60. doi: 10.1136/jech-2014-204708. Epub 2014 Nov 11. PMID 25389300
- [Derived] Ortega G, Castella C, Martin-Cantera C, Ballve JL, Diaz E, Saez M, Lozano J, Rofes L, Morera C, Barcelo A, Cabezas C, Pascual JA, Perez-Ortuno R, Salto E, Valverde A, Jane M; BIBE Study Group. Passive smoking in babies: the BIBE study (Brief Intervention in babies. Effectiveness). BMC Public Health. 2010 Dec 20;10:772. doi: 10.1186/1471-2458-10-772. PMID 21171981